CLINICAL TRIAL: NCT05342415
Title: Investigation of the Effect of Externally vs. Internally Focused Techniques on Thigh Muscle Activation After After Anterior Cruciate Ligament Reconstruction: A Randomized Assessor-Blinded Controlled Trial
Brief Title: Effect of Different Focused Techniques on Thigh Muscle Activation After Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dilara Kara, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FTREK24/31
Record Dates: First submitted 2022-04-03; First posted 2022-04-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: external focus; internal focus; knee rehabilitation; electromyography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The pre-and-post measurements will be performed by researchers who do not know the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internally Focused (Active Comparator): Focusing on the muscles that reveal the movement.
  Interventions: Other: Internally Focused Exercise
- Externally Focused (Experimental): Focusing on the result of the movement.
  Interventions: Other: Externally Focused Exercise

INTERVENTIONS:
Other: Internally Focused Exercise — While performing the exercises participants will be instructed to focus on the muscle itself.
  Arms: Internally Focused
Other: Externally Focused Exercise — While performing the exercises participants will be instructed to focus on the external target (towel, target line, etc.)
  Arms: Externally Focused

SUMMARY:
In recent years, it has been shown that different focuses (externally vs. internally focused) used when explaining exercises to patients after knee surgeries affect exercise performance and rehabilitation outcomes. Quadriceps muscle inhibition after anterior cruciate ligament reconstruction is one of the primary symptoms that should be treated. This study aimed to investigate the effects of different focusing techniques during the rehabilitation exercises after anterior cruciate ligament rehabilitation.

DETAILED DESCRIPTION:
Exercises are given for the symptoms of knee edema, knee range of motion, and quadriceps reflex inhibition in the acute period after anterior cruciate ligament surgery. In recent years it has been shown that the different focuses when explaining exercises to patients affect exercise performance and rehabilitation outcomes. It has been shown that the increase in performance of some exercises that require strength and power, such as long jump and sprint, especially with the applied external focus (the method of focusing on the result of the movement). However, it has been shown that there is an increase in muscle activation with internal focus (focusing on the muscles that reveal the movement). There is no study examining the effects of focusing differences on the exercise program given after anterior cruciate ligament reconstruction, especially on muscle activation after knee reflex inhibition.

30 individuals between the ages of 18-and 30 who had undergone anterior cruciate ligament reconstruction for the first time will be included in the study. The first evaluation will be performed and rehabilitation will begin in the first week after surgery. Patients who were taken into rehabilitation after anterior cruciate ligament surgery will be distributed into two different groups by the block randomization method. The same structured exercise program will be applied to the patients in both groups. Only the commands given during the exercise will be different.

Group 1: Internal Focused Exercise: E.g; While describing the knee pressing exercise (quadriceps isometric) in the long sitting position, the command "press your knee towards the bed by squeezing your thigh muscle" will be given by showing the muscle.

Group 2: External Focused Exercise: E.g; While describing the knee pressing (quadriceps isometric) exercise in the long sitting position, the command "press the towel/cloth that we put under your knee and compress your knee" will be given by showing the towel.

Patients will be followed under the supervision of a physiotherapist in the clinic 2 days a week and exercise progression will be provided. On the other days, the exercises will be continued as a home program. In order for the patients to comply with the exercises more easily and to be reminded easily, an exercise brochure will be given to the patients with the commands written and the exercises explained with pictures.

The last measurements will be performed at the end of one month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* who underwent anterior cruciate ligament reconstruction with hamstring tendon autograft for the first time
* no systemic inflammation
* agreed to participate in the study

Exclusion Criteria:

* having a chronic disease/injury in the ankle, hip and knee
* contralateral knee symptoms and/or surgery history
* other surgeries in addition to the anterior cruciate ligament reconstruction (meniscus repair, chondral surgery, etc.)
* post-operative referral of the patient more than a week later

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Determine if different focus techniques change thigh muscle activation | Baseline and 1 month after surgery
  Vastus medialis, vastus lateralis, and rectus femoris muscle activation will be measured by superficial electromyography

SECONDARY OUTCOMES:
Knee edema | Baseline and 1 month after surgery
  The changes in the limb circumference will be measured with a tape measure (cm).
Knee range of motion | Baseline and 1 month after surgery
  The changes in knee flexion and extension degree will be measured with a goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Volga Bayrakcı Tunay, PhD, Prof., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saka T. Principles of postoperative anterior cruciate ligament rehabilitation. World J Orthop. 2014 Sep 18;5(4):450-9. doi: 10.5312/wjo.v5.i4.450. eCollection 2014 Sep 18. PMID 25232521
- [Background] Kim DK, Hwang JH, Park WH. Effects of 4 weeks preoperative exercise on knee extensor strength after anterior cruciate ligament reconstruction. J Phys Ther Sci. 2015 Sep;27(9):2693-6. doi: 10.1589/jpts.27.2693. Epub 2015 Sep 30. PMID 26504270
- [Background] Cavanaugh JT, Powers M. ACL Rehabilitation Progression: Where Are We Now? Curr Rev Musculoskelet Med. 2017 Sep;10(3):289-296. doi: 10.1007/s12178-017-9426-3. PMID 28791612
- [Background] Sonnery-Cottet B, Saithna A, Quelard B, Daggett M, Borade A, Ouanezar H, Thaunat M, Blakeney WG. Arthrogenic muscle inhibition after ACL reconstruction: a scoping review of the efficacy of interventions. Br J Sports Med. 2019 Mar;53(5):289-298. doi: 10.1136/bjsports-2017-098401. Epub 2018 Sep 7. PMID 30194224
- [Background] Halperin I, Williams KJ, Martin DT, Chapman DW. The Effects of Attentional Focusing Instructions on Force Production During the Isometric Midthigh Pull. J Strength Cond Res. 2016 Apr;30(4):919-23. doi: 10.1519/JSC.0000000000001194. PMID 27003451
- [Background] Porter JM, Anton PM, Wikoff NM, Ostrowski JB. Instructing skilled athletes to focus their attention externally at greater distances enhances jumping performance. J Strength Cond Res. 2013 Aug;27(8):2073-8. doi: 10.1519/JSC.0b013e31827e1521. PMID 23222082
- [Background] Ille A, Selin I, Do MC, Thon B. Attentional focus effects on sprint start performance as a function of skill level. J Sports Sci. 2013;31(15):1705-12. doi: 10.1080/02640414.2013.797097. Epub 2013 May 28. PMID 23710928
- [Background] Marchant DC, Greig M, Scott C. Attentional focusing instructions influence force production and muscular activity during isokinetic elbow flexions. J Strength Cond Res. 2009 Nov;23(8):2358-66. doi: 10.1519/JSC.0b013e3181b8d1e5. PMID 19826287
- [Background] Schoenfeld BJ, Vigotsky A, Contreras B, Golden S, Alto A, Larson R, Winkelman N, Paoli A. Differential effects of attentional focus strategies during long-term resistance training. Eur J Sport Sci. 2018 Jun;18(5):705-712. doi: 10.1080/17461391.2018.1447020. Epub 2018 Mar 13. PMID 29533715
- [Background] Wulf G, Dufek JS, Lozano L, Pettigrew C. Increased jump height and reduced EMG activity with an external focus. Hum Mov Sci. 2010 Jun;29(3):440-8. doi: 10.1016/j.humov.2009.11.008. Epub 2010 Apr 21. PMID 20409600
- [Background] Kal EC, van der Kamp J, Houdijk H. External attentional focus enhances movement automatization: a comprehensive test of the constrained action hypothesis. Hum Mov Sci. 2013 Aug;32(4):527-39. doi: 10.1016/j.humov.2013.04.001. Epub 2013 Jun 30. PMID 24054892
- [Background] Ogrodzka-Ciechanowicz K, Glab G, Slusarski J, Gadek A. Quadriceps muscle strength recovery with the use of high tone power therapy after anterior cruciate ligament reconstruction: a randomized controlled trial. BMC Musculoskelet Disord. 2021 Nov 23;22(1):975. doi: 10.1186/s12891-021-04862-w. PMID 34814896